CLINICAL TRIAL: NCT04559152
Title: Zinc Supplementation During Pregnancy for the Prevention of Stunting: Analysis of Maternal Serum Zinc, Cord Blood Osteocalcin and Neonatal Birth Length
Brief Title: Zinc Supplementation During Pregnancy: Analysis of Maternal Serum Zinc, Cord Blood Osteocalcin and Neonatal Birth Length
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitas Sumatera Utara (Other)
Responsible Party: Principal Investigator, Lili Rohmawati, Zinc Supplementation During Pregnancy for the Prevention of Stunting: Analysis of Maternal Serum Zinc, Cord Blood Osteocalcin and Neonatal Birth Length, Universitas Sumatera Utara
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 9/UN5.2.3.1/PPM/KP-DRPM/2019
Record Dates: First submitted 2020-09-09; First posted 2020-09-22 (Actual); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Zinc Deficiency; Birth Length
Keywords: Zinc; Maternal zinc; Osteocalcin; Birth length

STUDY DESIGN:
Intervention Model Description: An experimental study with pre-test/post-test control groups, double-blind with randomization block technique
Who Masked: Participant, Investigator
Masking Description: The subjects were divided into two groups (zinc supplementation and a placebo (control) group). Researchers and the subjects did not know the type of zinc supplementation or placebo given. The blinding process is carried out by the research assistant to the subject in the field at the time of retrieval of the research data. The selection of samples for each group uses the blocked randomization technique.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Zinc Supplementation Group (Experimental): Zinc capsule (20mg) was taken in the morning after meals once daily for 12 weeks. All subjects in this arm were also given iron and folic acid tablets in accordance with the Indonesian government program.
  Interventions: Dietary Supplement: Zinc Supplementation Group
- Placebo Group (Placebo Comparator): Placebo (sugar tablet) was taken in the morning after meals once daily for 12 weeks. All subjects were also given iron and folic acid tablets in accordance with the Indonesian government program. Each placebo tablet was inserted into a capsule of the same shape and color with zinc capsule
  Interventions: Dietary Supplement: Placebo Group

INTERVENTIONS:
Dietary Supplement: Zinc Supplementation Group — Enrolled subjects received zinc capsule 20mg daily in the morning after meal for 12 weeks
  Arms: Zinc Supplementation Group
Dietary Supplement: Placebo Group — Enrolled subjects received placebo tablet, which was inserted into capsule of the same shape and color as zinc capsule, daily in the morning after meal for 12 weeks
  Arms: Placebo Group

SUMMARY:
This experimental study was conducted with pre-test/post-test control groups and double-blind randomization from March to December 2019 at Universitas Sumatera Utara Hospital and others in Medan. Subjects were pregnant mothers in second or third trimester and with their newborns who met the inclusion criteria. Subjects were divided into two groups and administered either zinc supplementation 20 mg/day or placebo, respectively, for 12 weeks. The parameters assessed were maternal serum zinc levels cord blood osteocalcin and birth length measurements.

DETAILED DESCRIPTION:
Patients and Study Design This was an experimental study with pre-test/post-test control groups, double-blind with randomization block technique. This study was conducted from March to December 2019 in the obstetrics and neonatology unit of Universitas Sumatera Utara Hospital, Malahayati Islamic Hospital and Royal Maternity Hospital in Medan. Research subjects were pregnant mothers with their newborns who met the inclusion criteria. The study samples were divided into two groups and administered either zinc supplementation 20 mg/day or placebos, respectively, for 12 weeks. The zinc tablets or placebos were given in the morning after meals. All subjects were also given iron and folic acid tablets in accordance with the Indonesian government program. Subjects were healthy pregnant mothers in their second or third trimester, 20-35 years old, with a height of >150 cm and no indication of cons following this study, as determined by obstetrician and gynaecology specialists; subjects were enrolled with a consecutive sampling technique. Births involving twins, congenital abnormalities, prematurity (gestation age <37 weeks) or stillbirth were excluded.

Informed consent was given by all subjects' legal guardians following the provision of sufficient information prior to the study.

This study was approved by the Health Research Ethical Committee, School of Medicine, Universitas Sumatera Utara in accordance with the principles of the Helsinki Declaration (No.179/TGL/FK USU-RSUP HAM/2019).

Methods The parameters assessed in this study were maternal serum zinc levels, cord blood osteocalcin and birth length measurements. Maternal serum zinc levels were measured twice with 6 ml of vein blood each time, both during initial antenatal care and after 12 weeks of supplementation. Samples were subsequently centrifuged for 15 minutes at 3000 rpm. Specimens were processed by the inductively coupled plasma-mass spectrometry (ICP-MS) method using Agilent 7700 analyser (Santa Clara, USA, 2014). Normal serum zinc levels were defined based on a cut-off value of ≥ 56 µg/dL in accordance with Second National Health and Nutrition Examination Survey data from 1976-1980 (NHANES II).

Cord blood osteocalcin levels were measured with 6 ml cord blood samples prior to delivery, which were subsequently centrifuged for 15 minutes at 1000 rpm using Cobas e601 analyser (Roche Diagnostic, Mannheim, Germany) and N-Mid Osteocalcin (Abbexa) reagent. Osteocalcin was measured using the enzyme-linked immuno-sorbent assay (ELISA) method, and in accordance with Prodia clinical laboratory standards.

Neonatal birth length was performed with a SECA 232 digital baby scale for length with an accuracy of 0.1 cm. Maternal zinc intake was calculated in accordance with the NutriSurvey 2007 Indonesian version.

Statistical Analysis Descriptive analyses, correlation tests, and linear regression tests were performed using SPSS version 23.0 (SPSS Inc., Chicago, Illinois, USA). Statistical significance was considered at a p-value < 0.05 with a 95% confidence interval.

ELIGIBILITY:
Inclusion Criteria:

* Healthy pregnant mothers in their second or third trimester
* Age 20-35 years old
* Minimal height 150 cm

Exclusion Criteria:

Pregnant mothers in high-risk conditions such as

* severe malnutrition
* eclampsia
* gestational diabetes
* liver diseases
* kidney diseases

Neonatal with

* twin babies
* congenital anomalies
* prematurity (gestation age <37 weeks)
* stillbirth

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant mothers and their newborn babies
Enrollment: 71 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Zinc Supplementation During Pregnancy Prevent Stunting Occurence to the Newborn: Analysis of Maternal Serum Zinc, Cord Blood Osteocalcin and Neonatal Birth Length | 12 weeks up to childbirth
  Maternal serum zinc level (after intervention) was measured and analysed statistically for its correlation with mean cord blood osteocalcin levels and median neonatal birth lengths

SECONDARY OUTCOMES:
Correlation Between Maternal Zinc Supplementation with Maternal Serum Zinc Levels | 12 weeks
  Maternal Serum Zinc level was measured before and after intervention. Participants dietary intake also will be accounted and calculated via food recall.
  The serum zinc level before and after intervention will then be analysed statistically to check for any correlation between zinc dietary intake and serum zinc level

CONTACTS AND LOCATIONS:
Overall Officials: Lili Rohmawati, Researcher, Principal Investigator — Universitas Sumatera Utara
Locations (1):
- Universitas Sumatera Utara, Medan, North Sumatra, Indonesia

IPD SHARING:
Plan to Share IPD: Yes
The results of this study
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Agustus 2020
Access Criteria: lily_rahmawati234@yahoo.com

REFERENCES:
- [Result] Rohmawati L, Keumala DS, Sitepu M. Maternal Zinc Intake and Its Correlation with Maternal Serum Zinc Levels and Neonatal Birth Weight/Length. Pak. J. Nutr., 19 (5): 245-252, 2020. DOI: 10.3923/pjn.2020.245.252